CLINICAL TRIAL: NCT00661986
Title: Effect of Different Dosages of Dark Chocolate on Arterial Blood Pressure in Cardiovascular High-risk Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Leipzig (Other)
Responsible Party: Steffen Desch, University of Leipzig
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Leipzig chocolate
Record Dates: First submitted 2008-04-17; First posted 2008-04-21 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2010-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): dark chocolate 6 g/day
  Interventions: Dietary Supplement: dark chocolate 6 g/day
- 2 (Active Comparator): dark chocolate 25 g/day
  Interventions: Dietary Supplement: dark chocolate 25 g/day

INTERVENTIONS:
Dietary Supplement: dark chocolate 6 g/day — dark chocolate 6 g/day
  Arms: 1
Dietary Supplement: dark chocolate 25 g/day — dark chocolate 25 g/day
  Arms: 2

SUMMARY:
Low habitual intake of low-dose dark chocolate (6 g/day) has been shown to have a beneficial effect on arterial blood pressure in one previous study. The trial will assess if ingestion of a higher but still moderate dose (25 g/day) over 3 months will have a more pronounced effect. The population will consist of cardiovascular high-risk patients only (who will potentially benefit most from blood-pressure lowering).

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* mean ambulatory blood pressure 125-146 mmHg and/or 80-89 mmHg
* high cardiovascular risk profile (one or more of the following: CAD, PAD, carotid stenosis, diabetes)
* informed consent

Exclusion Criteria:

* habituary intake of dark chocolate or cocoa products
* mean ambulatory blood pressure 147 mmHg or greater and/or 90 mmHg or greater
* pregnancy
* uncontrolled diabetes
* severe comorbidity
* change in blood pressure medication within last 6 weeks
* participation in another trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2008-02; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
change in mean ambulatory arterial blood pressure | 3 months

SECONDARY OUTCOMES:
change in weight and BMI | 3 months
change in various lab parameters | 3 months